CLINICAL TRIAL: NCT00577057
Title: Randomized Trial to Evaluate the Therapeutic Gain by Changing the Chemoradiotherapy From Concurrent-adjuvant to Induction-concurrent Sequence, and the Radiotherapy From Conventional to Accelerated Fractionation for Advanced Nasopharyngeal Carcinoma
Brief Title: Benefit of Changing Chemoradiotherapy Sequence and Modifying Radiotherapy Schedule for Advanced Nasopharyngeal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: Hong Kong Nasopharyngeal Cancer Study Group Limited (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: HKEC-2006-120; HARECCTR0500062; NPC-0501
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Nasopharyngeal Neoplasms
Keywords: Nasopharyngeal Carcinoma; Stage III - IVB
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Nasopharyngeal Carcinoma | interventions — Cisplatin; Fluorouracil; Capecitabine

INTERVENTIONS:
Procedure: Conventional Radiotherapy
Procedure: Accelerated Radiotherapy
Drug: Cisplatin
Drug: 5-fluorouracil
Drug: Capecitabine

SUMMARY:
The objectives of this clinical study are threefold:

1. To compare the benefits in cancer control and survival obtained from adding induction-concurrent chemotherapy to radiation with those from adding concurrent-adjuvant chemotherapy to radiation.
2. To test whether replacing fluorouracil with Xeloda in combining with cisplatin (PF or PX, respectively) in the chemotherapy plan will maintain or improve further the chemotherapy benefits while reducing the duration of hospital stay.
3. To see if accelerated fractionation radiotherapy can improve the outcome of patients as compared with conventional fractionation radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven nasopharyngeal carcinoma
* Non-keratinizing or undifferentiated type Stage III-IVB (by AJCC/UICC 6th edition)
* Essential staging investigations: CT or MRI of nasopharyngeal region Chest x-ray (or CT thorax)
* Liver function test, alkaline phosphatase Liver and bone scan if alkaline phosphatase exceeds the institutional upper limit of normal, or if clinically indicated.
* Liver scan if SGOT exceeds the institutional upper limit of normal
* Adequate marrow: WBC > 4 and platelet > 100
* Adequate renal function: creatinine clearance > 60 ml/min.
* Satisfactory performance status: > 2 by ECOG System.

Exclusion Criteria:

* WHO Type I squamous cell carcinoma or adenocarcinoma
* Age > 70
* Treatment with palliative intent (including those with tumor extent mandating the use of AP opposing facio-cervical field technique)
* Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in-situ cervical cancer, or other cancer for which the patient has been disease-free for five years.
* Pregnancy or lactation (consider pregnancy test in women of child-bearing age and emphasize effective contraception during the treatment period).
* History of previous RT (except for non-melanomatous skin cancers outside intended RT treatment volume).
* Prior chemotherapy or surgery (except diagnostic) to primary tumor or nodes.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 798 (Estimated)
Dates: Start 2006-09; Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 5-year
Overall Survival | 5-year

SECONDARY OUTCOMES:
Overall / Locoregional / Distant Failure Free Rate | 5-year
Chemotherapy and RT toxicity | within 90 day from commencement of RT
Late Toxicity | 5-year

CONTACTS AND LOCATIONS:
Overall Officials: Anne WM Lee, Cos, Principal Investigator — Clinical Oncology, Pamela Youde Nethersole Eastern Hospital
Locations (6):
- China (6):
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - Prince of Wales Hospital, Hong Kong
  - Princess Margaret Hospital, Hong Kong
  - Queen Elizabeth Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Tuen Mun Hospital, Hong Kong